CLINICAL TRIAL: NCT04441489
Title: Assessment of Lung Inflammation With FDG PET/CT in COVID-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: PET-COVID
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; FDG PET/CT; Inflammation
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to assess the inflammatory status at the presumed peak of the inflammatory phase in non-critically ill patients requiring admission for COVID-19. Patients admitted with COVID-19 from March 27th to May 3rd, 2020 were prospectively enrolled. All patients had an initial chest CT-scan for diagnosis on admission and a second chest CT-scan for follow-up concomitant with a FDG PET/CT between day 6 and day 14 after the onset of symptoms.

DETAILED DESCRIPTION:
[18F]-2-fluoro-2-deoxy-D-glucose PET/CT (FDG PET/CT) is a sensitive and quantitative technic for detecting inflammatory process. Glucose uptake is correlated with increased anaerobic glycolysis seen in activated inflammatory cells such as monocytes, lymphocytes and granulocytes.

The aim of the study was to assess the inflammatory status at the presumed peak of the inflammatory phase in non-critically ill patients requiring admission for COVID-19.

Patients were included if COVID-19 was confirmed according to the WHO guidance (11) by a positive result of RT-PCR assay of nasal and pharyngeal swabs, if they were hospitalized during the time period from day 6 to day 14 of the onset of symptoms, and if their initial (on admission) chest CT-scan presented ground-glass opacities (GGO) or consolidation.

Group of 13 consecutive patients prospectively enrolled. All patients had an initial chest CT-scan for diagnosis on admission and a second chest CT-scan for follow-up concomitant with a FDG PET/CT between day 6 and day 14 after the onset of symptoms.

Based on the changes between the two chest CT, patients were classified as follows:

* CT worsening: increase of CT abnormalities extent > 20% or additional GGO or consolidation. Conversion of GGO into consolidation was not considered as additional finding.
* CT stability: changes of CT abnormalities extent ≤ 20% without additional GGO or consolidation.
* CT improvement: decrease of CT abnormalities extent > 20% without additional GGO or consolidation.

Based on FDG PET/CT imaging, patients' profiles were classified as follows:

* Inflammatory: lungs hypermetabolic volume ≥ 50 ml and / or SUVmax ≥ 7
* Low inflammatory: lungs hypermetabolic volume < 50 ml and / or SUVmax< 7 Patients' short-term clinical outcome was classified as follows: worsening, stability, improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if COVID-19 was confirmed according to the WHO guidance (11) by a positive result of RT-PCR assay of nasal and pharyngeal swabs, if they were hospitalized during the time period from day 6 to day 14 of the onset of symptoms, and if their initial (on admission) chest CT-scan presented ground-glass opacities (GGO) or consolidation.

Exclusion Criteria:

* Patients could not be included if their medical condition was unstable or precluded a safe transfer to the nuclear medicine department, if they were under mechanical ventilation (either non-invasive or invasive), if they were initially referred to the critical care unit, and in case of a pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with COVID-19 from March 27th to May 3rd, 2020 were prospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | Day 6 to Day 14
  Amount of FDG pathological uptake expressed by maximum signal intensity standardized uptake values (SUVmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Derived] Dietz M, Chironi G, Claessens YE, Farhad RL, Rouquette I, Serrano B, Nataf V, Hugonnet F, Paulmier B, Berthier F, Keita-Perse O, Giammarile F, Perrin C, Faraggi M; MONACOVID Group. COVID-19 pneumonia: relationship between inflammation assessed by whole-body FDG PET/CT and short-term clinical outcome. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):260-268. doi: 10.1007/s00259-020-04968-8. Epub 2020 Jul 25. PMID 32712702